CLINICAL TRIAL: NCT04346576
Title: The Effects of Fermented Milk Including Lactobacillus Casei Strain Shirota Regarding Gastrointestinal Symptoms, Respiratory Infection, Nutrition Improving in Vietnam Children 3-5 Years of Age
Brief Title: Probiotics Prevent Health Problems in Children
Acronym: Shirota
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Institute of Nutrition, Vietnam (Other Government)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Principal Investigator, TRUONG TUYET MAI, Associate Professor, PhD, MD, National Institute of Nutrition, Vietnam
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: NINVN12017; R01DA013131 (NIH)
Record Dates: First submitted 2020-03-29; First posted 2020-04-15 (Actual); Last update posted 2020-04-15 (Actual); Status verified 2020-04

CONDITIONS: Gastrointestinal System Disease; Respiratory System
Keywords: Lactobacillus casei strain Shirota; diarrhea, constipation; respiratory system; nutrition status; children 3-5 years old
MeSH Terms: conditions — Digestive System Diseases; Diarrhea; Constipation

STUDY DESIGN:
Intervention Model Description: A controlled field trial was implemented with 1,036 children (3-5 years old) in Thanh Hoa province in Vietnam. The probiotic group (n=518) consumed 65 mL/day of fermented milk containing 108 CFU/mL of LcS for the 12-week intervention period, whereas the control group did not. The incidence of constipation, diarrhea, ARI, and anthropometry in children was determined at baseline and 4, 8, and 12-week of intervention and after the 4-week follow up period.
Masking Description: A controlled field trial was implemented with 1,036 children (3-5 years old) in Thanh Hoa province in Vietnam. The probiotic group (n=518) consumed 65 mL/day of fermented milk containing 108 CFU/mL of LcS for the 12-week intervention period, whereas the control group did not. The incidence of constipation, diarrhea, ARI, and anthropometry in children was determined at baseline and 4, 8, and 12-week of intervention and after the 4-week follow up period.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Probiotics (LcS per 65 mL) prevent health problems in children (Experimental): Probiotic test product was fermented milk containing 6.5 billion of LcS per 65 mL (108 CFU/mL), manufactured by Yakult Vietnam, Co., Ltd. The nutritional composition of the test product is 0.8 g of protein, <0.1 g of fat, 12.4 g of carbohydrates, and the total energy is 52.7 kcal per bottle. Subjects were asked to drink one bottle of the test product per day after lunch for 12 weeks on consecutive days. The test products were stored in a refrigerator (< 10°C), protected from direct sunlight, and used before their expiration date. Adherence to the intervention protocol was confirmed as follows; teachers at kindergartens or parents at home provided the probiotic drinks (1 bottle/day x 7 days/week) after lunch.
  Interventions: Dietary Supplement: Probiotics prevent health problems in children

INTERVENTIONS:
Dietary Supplement: Probiotics prevent health problems in children — A controlled field trial was conducted with 1,036 children (3-5 years old) in Thanh Hoa province in Vietnam. The probiotic group (n=518) consumed fermented milk 65 mL/day containing 108 CFU/mL of LcS for the 12-week intervention period, whereas the control group (n=493) were not given any. The incidence of constipation, diarrhea, ARI, and anthropometry in children was determined at baseline, after 4, 8, and 12-week intervention and after the 4-week follow-up period.
  Other Names: Yakult fermented milk

SUMMARY:
Randomized controlled field trial of a probiotics to assess its roles in the prevention or improvement of constipation and diarrhea, acute respiratory infection, nutrition improving in Vietnam children.

In the present proposal, the investigators plan to examine if daily intake of a probiotic beverage, which includes 6.5 billion probiotic Lactobacilli, has a beneficial role in protecting children from infectious diarrhea and constipation in Vietnam with 3 objectives:

1. To assess the impact of probiotics in the prevention or improvement of diarrhea and constipation in children
2. To assess the impact of probiotics in the prevention of disease of respiratory system (ARI)
3. To assess the impact of probiotics on nutrition and growth of the children

DETAILED DESCRIPTION:
It will be a randomized controlled field trial involving 1036 children aged between 3 and 5 years in some communities in Vietnam. The 1036 children will be identified through demographic survey. Based on available National data to determine the province - Thanh Hoa province (http://viendinhduong.vn/news/vi/106/61/0/a/so-lieu-thong-ke-ve-tinh-trang-dinh-duong-tre-em-qua-cac-nam.aspx), after surveying 2.000 children at least 6 communes, it is expected to give 1036 eligible children. The study will be randomized where the treatment group will receive Probiotic drink, which includes 65 billion probiotic Lactobacillus casei strain Shirota, one bottle (65ml) daily for 12 weeks and the non-treatment arm will not receive the probiotic drink for 12 weeks. Randomization will be done in a ratio of 1:1, i.e., the study arm and control arm will include 518 children each. All the children under the study will be visited daily by a by teachers at kindergartens (when the children attend class), or by parents (when the children are at home). The surveillance persons will supervise the intake of Probiotic drink by the children, the status of diarrhea and constipation, disease of respiratory in children and recording the data every day. All the children will be followed up daily for 4 weeks (after stop the intervention) for identification of diarrhea and constipation cases. Functional constipation defined by ROME III was evaluated every 4 weeks. It was diagnosed by doctors with reference to the logbook records. The stool consistency was recorded in a daily logbook based on the Bristol Stool Form Scale. Diarrhea will be defined as three or more abnormally loose or liquid stools within last 24 h period. Details of such diarrhea cases including their duration, frequency of stool, type of stool (watery or bloody), other associated symptoms like abdominal pain etc. will be recorded. Qualified medical doctors will provide services for appropriate counseling and treatment and severe cases will be referred to the hospital. Doctors at commune stations are collaborate to provide service for appropriate counseling and treatment during the time of trial. And doctors at district hospitals and Thanh Hoa province will be collaborated to treat with severe cases when they are referred to. Measurements of height, weight and mid-arm circumference will assess nutritional status of the children at the beginning of the study, at the end of 4, 8, 12 weeks and (at the end of 16 weeks) follow up for 4 weeks. The outcome variables will be the incidence of diarrhea, constipation, disease of respiratory, nutrition status and the efficacy of the probiotics will be calculated by comparing the diarrhea, constipation incidence, disease of respiratory between the two groups at 5 different point of time (at baseline, the end of 4, 8, 12 weeks and 16 weeks). Nutritional improving will be compared similarly at baseline, the end of 4, 8, 12 weeks and 16 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Children of either sex aged 3-5 years who are attending the school
* The parents/ guardians of each participating child agreed in their child participant and signed the consent form.

Exclusion Criteria:

* Children with Alzheimer's disease
* Children using long-term antibiotics
* Children with inborn chronic disease such as congenital heart disease; congenital chronic kidney failure.
* Two children in the same home (the same parents)

Ages: 3 Years to 5 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Gender Based: Yes — The list of children was identified in the school, including female and male
Enrollment: 1036 (Actual)
Dates: Start 2017-10-05 (Actual); Primary Completion 2018-01-05 (Actual); Study Completion 2018-06-05 (Actual)

PRIMARY OUTCOMES:
Incidence of constipation disease | 16 weeks (12 weeks of intervention and 4-weeks follow-up)
  In the primary analysis, the denominator in the calculation of incidence of constipation disease (/100 children/ week) will consist of the number of eligible children living in the study area at the time of the trial who were in between 3-5 year of age. Individuals will be included in the denominator until out-migration, death. All children will be included in the corresponding group during analyses.
Incidence of respiratory (ARI) | 16 weeks (12 weeks of intervention and 4-weeks follow-up)
  In the primary analysis, the denominator in the calculation of incidence (/100 children/ week) will consist of the number of eligible children living in the study area at the time of the trial who were in between 3-5 year of age. Individuals will be included in the denominator until out-migration, death. All children will be included in the corresponding group during analyses.
Average duration of diarrhea | 16 weeks (12 weeks of intervention and 4-weeks follow-up)
  Average duration of diarrhea were calculated during 12 weeks of intervention period and 4 weeks of follow-up period. If there are at least 3 diarrhea-free days between a first and a second episode of diarrhea in the same individual, the second diarrhea episode were considered as a separate (new) diarrheal episode. Evaluation of probiotic efficacy thus pertains to number of diarrheal episodes. Average duration of diarrhea were average of the day number of episodes that were determined.
Incidence of diarrhea disease | 16 weeks (12 weeks of intervention and 4-weeks follow-up)
  n the primary analysis, the denominator in the calculation of incidence of diarrhea disease (/100 children/ week) will consist of the number of eligible children living in the study area at the time of the trial who were in between 3-5 year of age. Individuals will be included in the denominator until out-migration, death. All children will be included in the corresponding group during analyses.
Average duration of constipation | 16 weeks (12 weeks of intervention and 4-weeks follow-up)
  Average duration of constipation were calculated during 12 weeks of intervention period and 4 weeks of follow-up period. The diagnosed constipation days between a first and a second episode of constipation in the same individual, the second constipation episode were considered as a separate (new) constipation episode. Evaluation of probiotic efficacy thus pertains to number of constipation episodes. Average duration of constipation were average of the day number of episodes that were determined.
Average duration of ARI | 16 weeks (12 weeks of intervention and 4-weeks follow-up)
  Average duration of ARI were calculated during 12 weeks of intervention period and 4 weeks of follow-up period. The diagnosed ARI days between a first and a second episode of ARI in the same individual, the second ARI episode were considered as a separate (new) ARI episode. Evaluation of probiotic efficacy thus pertains to number of ARI episodes. Average duration of ARI were average of the day number of episodes that were determined.
The weight gain | 16 weeks (12 weeks of intervention and 4-weeks follow-up)
  Using TANITA electronic scales with accuracy up to 0.1 kg determine the weight of children.
  The weight gain were determined the weight change of children after intervention compared of that before intervention. These weight gain were compared among the treatment and non-treatment group.
The height gain | 16 weeks (12 weeks of intervention and 4-weeks follow-up)
  The height was measured by the vertical height meter with accuracy up to 1 mm. The height gain were determined the height change of children after intervention compared of that before intervention. These height gain were compared among the treatment and non-treatment group.
The changes in the Z-score | 16 weeks (12 weeks of intervention and 4-weeks follow-up)
  Assess the nutritional status of children based on Z-Score (WHO-2006). The change in Zscore were compared among the treatment and non-treatment group.

SECONDARY OUTCOMES:
Dietary intake | 16 weeks (12 weeks of intervention and 4-weeks follow-up)
  Using 24 hours recall to do the dietary intake

CONTACTS AND LOCATIONS:
Overall Officials: Tuyen Le, Study Director — National Institute of Nutrition
Locations (1):
- Cong Chinh, Van Thang, Dinh Thanh and Yen Thai, Thanh Hóa, Thanh Hóa Province, Vietnam

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Informed Consent Form (2017-09-15): https://cdn.clinicaltrials.gov/large-docs/76/NCT04346576/ICF_000.pdf